CLINICAL TRIAL: NCT00989443
Title: A Phase I Clinical Study to Evaluate the Tolerance and Safety of an Aqueous Gel Containing 2% (w/w) of Cidofovir, Directly Applied on the Cervix Exhibiting High Grade Squamous Intraepithelial Lesion(s) (CIN 2 and 3)
Brief Title: Safety and Tolerability of Cidofovir Gel Applied on Cervix Squamous Lesions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mithra Pharmaceuticals (Industry)
Responsible Party: Dr. Michel Bossens, Erasme Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-COL-CI01; EudraCT2009-012937-31
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Uterine Cervical Neoplasms; Cervix Intraepithelial Neoplasia
Keywords: Cervix Intraepithelial Neoplasia grades 2 and 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cidofovir (Experimental)
  Interventions: Drug: Cidofovir gel

INTERVENTIONS:
Drug: Cidofovir gel — topical gel applied once a week for 3 weeks

SUMMARY:
Human Papilloma Virus (HPV) infections induce cervical intraepithelial neoplasia (CIN) of cervix. To reduce incidence of invasive tumor associated with high grade CIN lesions, the standard treatment is the conisation of cervix (surgical act). A local treatment with the antiviral and anti-proliferative cidofovir would preserve the cervix of young subjects and reduce obstetrical morbidity induced by the conisation.

This clinical study is aimed at :

1. evaluating the tolerance and safety of a cidofovir gel directly applied on the cervix exhibiting high grade CIN lesions;
2. evaluating the pharmacokinetic (PK) profile of cidofovir after local application.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 18 and 50 years old
* volunteers
* informed consent signed
* cervical lesion classified CIN 2 or 3, on a biopsy made during the 6 preceding weeks
* no sexual activity or use of effective mechanical, hormonal or intrauterine contraception (except hormonal vaginal ring)

Exclusion Criteria:

* pregnancy or breast feeding
* subtotal hysterectomy
* current or ancient renal impairment
* current immune disorder
* current use of drugs interfering with renal function
* current treatment for any cancer
* current use of treatment interfering with immunity
* current use of anti-viral treatment
* current or recent participation to another experimental study during the last 3 months before the screening visit
* current vaginal application of drugs or cosmetics
* local or general condition incompatible with the experimental treatment in the opinion of the principal investigator

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
adverse events | weeks 1, 2, 3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Michel Bossens, MD, PhD, Principal Investigator — Erasme Hospital - Laboratoire de recherche en reproduction humaine
Locations (1):
- Erasme Hospital, Brussels, Belgium